CLINICAL TRIAL: NCT00549874
Title: Effect of Rosiglitazone on Myocardial Blood Flow Regulation in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SKB 276
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Last update posted 2007-11-09 (Estimated); Status verified 2007-10

CONDITIONS: Type 2 Diabetes
Keywords: insulin resistance; type 2 diabetes; myocardial perfusion; nitrosative stress; thiazolidinediones
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Rosiglitazone; Glyburide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Rosiglitazone
- 2 (Experimental)
  Interventions: Drug: Glyburide

INTERVENTIONS:
Drug: Rosiglitazone — oral 8 mg/once daily for 6 months
  Arms: 1
Drug: Glyburide — 20 mg/ once daily for 6 months
  Arms: 2

SUMMARY:
The overall hypothesis to be tested is that increased insulin resistance contributes to abnormal cardiac blood flow regulation in type 2 diabetic patients, which can be reversed by 6 months treatment with rosiglitazone. The planned experimental approach will be to utilize nuclear medicine techniques to evaluate whether the administration of rosiglitazone for 6 months can reverse regional deficits in myocardial blood flow and glucose utilization in type 2 diabetes in a randomized double blind controlled study. These studies will help elucidate the potential of rosiglitazone to correct deficits of myocardial blood flow complicating diabetes with the overall aim being the eventual prevention of sudden cardiac death.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* 30-75 years of age
* less than 1% fluctuation in HbA1c over 3 months
* women must be on contraception
* HbA1c 6-9%
* willingness to sign approved consent form

Exclusion Criteria:

* Nursing mothers, pregnant women (excluded by a negative pregnancy test).
* Subjects requiring insulin therapy (>20 units/day) and can not be converted to sulfonylurea therapy without loss of diabetes control.
* Patients with a history of drug or alcohol dependence in the last 5 years
* Patients with pre-existing cardiovascular disease including coronary artery disease, heart attack, heart failure, abnormal heart rhythms, structural abnormalities and valve disease, peripheral vascular disease and uncontrolled high blood pressure.
* Patients with a history of high cholesterol requiring therapy.
* Patients with severe systemic disease other than diabetes which has as a recognized complication neuropathy
* Patients currently taking drugs which act on the blood vessels (for example for hypertension)
* Patients taking antidepressants, or other drugs or medications known to interfere with the uptake or metabolism of catecholamines (stress hormones)
* Patients with poor renal function or have significant liver disease
* Patients with a history of previous kidney, pancreas or cardiac transplantation.
* Patients with a history of "severe hypoglycemia" which required the assistance of a third party or ketoacidosis requiring hospital admission within the last 3 months.
* Patients with lung disease for example resulting from chronic obstructive airways disease.
* Patients with abnormal thyroid function tests.
* Patients having taken other systemic investigational drugs (especially for neuropathy) or initiating a new or experimental insulin delivery device within 3 months of starting the study.
* Patients with a history of allergic reactions to multiple drugs or biological products.
* Obese patients (BMI greater than 35).
* Patients who refuse to sign the informed consent.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2002-02; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Myocardial blood flow regulation | 6 months intervention

SECONDARY OUTCOMES:
biomarkers of oxidative/nitrosative stress | 6 month intervention

CONTACTS AND LOCATIONS:
Overall Officials: Martin Stevens, MD, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - University of Toledo - Health Campus, Toledo, Ohio

REFERENCES:
- [Derived] Pop-Busui R, Oral E, Raffel D, Byun J, Bajirovic V, Vivekanandan-Giri A, Kellogg A, Pennathur S, Stevens MJ. Impact of rosiglitazone and glyburide on nitrosative stress and myocardial blood flow regulation in type 2 diabetes mellitus. Metabolism. 2009 Jul;58(7):989-94. doi: 10.1016/j.metabol.2009.02.020. PMID 19394661